CLINICAL TRIAL: NCT03418792
Title: Functional Sparing of Salivary Glands Using MRI Sialography for Patients Undergoing Definitive Radiation Therapy for Head and Neck Cancers of the Oropharynx
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LCCC 1735
Record Dates: First submitted 2018-01-25; First posted 2018-02-01 (Actual); Last update posted 2023-05-31 (Actual); Status verified 2023-05

CONDITIONS: Head and Neck Cancer; Oropharynx Cancer; Xerostomia Due to Radiotherapy
MeSH Terms: conditions — Head and Neck Neoplasms; Oropharyngeal Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Parotid-Sparing Head & Neck Radiation (Experimental): Patients with Oropharyngeal Squamous Cell Carcinoma (OPSCC) who will be treated with parotid-sparing head & neck radiation. MRI Sialograms will be obtained to identify salivary ductal structures and stem cells to be spared during treatment.
  Interventions: Other: Parotid-Sparing Head & Neck Radiation Guided by MRI Sialography

INTERVENTIONS:
Other: Parotid-Sparing Head & Neck Radiation Guided by MRI Sialography — Head & neck radiation with parotid sparing. Parotid sparing will be facilitated by avoidance of salivary ductal structures and stem cells, as identified by the pre-treatment MRI sialogram, in the radiation treatment plan.

SUMMARY:
The proposed study is an attempt to improve patient xerostomia (dry mouth) after definitive radiation therapy treatment for head and neck cancer. Xerostomia is a frequently experienced symptom for those receiving radiation therapies to the head and neck that persists after treatment, potentially indefinitely. It has been shown that stem/progenitor cells preferentially reside in large ducts of salivary glands and that these cells have the ability to repair radiation induced salivary damage. Current practice does not specifically attempt to spare these regions and considers the entire salivary gland to have equal importance and function. This study will involve the acquisition of pre-treatment MRI sialogram images which enable visualization of salivary ducts (using saliva itself as a contrast agent) that can then be avoided during radiation treatment planning. Saliva samples will also be collected at this time to quantify baseline saliva secretion and saliva characteristics. The primary objective will be to obtain patient reported outcomes (PRO) measure of xerostomia related symptoms for comparison with a historical cohort. Xerostomia symptom information will be obtained by use of a patient reported quality of life survey administered prior to treatment and at 6, 12, 18, and 24 months after treatment. The secondary objectives will be to quantitatively assess post-treatment changes in saliva secretion, salivary gland volume, and ductal visibility using MRI sialograms. The target sample size for this study is 40 patients. The investigator hypothesizes that reducing the dose to these stem cell containing salivary ducts will facilitate improvements in patient reported symptoms as well as improved recovery of salivary secretion, salivary gland volume, and intra-glandular ductal visibility using MRI sialograms.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* T0-4, N0-3, M0 disease of the oropharynx
* Will be treated with intensity modulated radiation therapy (IMRT) and with definitive intent (either definitive or postoperative radiotherapy)
* No contraindications to receiving an magnetic resonance imaging (MRI) such as: implanted electrical devices, pregnancy, and/or significant quantities of metal in the head/neck
* Radiologic confirmation of the absence of hematogenous metastasis within 12 weeks prior to treatment; at a minimum, chest x-ray is required (computerized tomography (CT) imaging of the chest or positron emission tomography (PET) /CT is acceptable)
* Eastern Cooperative Oncology Group (ECOG) Performance Status 0-2
* Able to comply with the treatment plan and follow-up schedule
* Provides study-specific informed consent prior to study entry

Exclusion Criteria:

* Sjogren's syndrome or baseline xerostomia (CTCAE > 0 for question regarding dry mouth)
* Lesions grossly involving the salivary glands
* Allergy to lemon juice
* Prior history of radiation therapy to the head and neck
* Pre-treatment scan deemed not usable

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-03-08 (Actual); Primary Completion 2022-04-22 (Actual); Study Completion 2023-05-02 (Actual)

PRIMARY OUTCOMES:
Xerostomia | One year after completion of IMRT on last enrolled patient
  Patient reported xerostomia (dry mouth) after IMRT with salivary ductal sparing

SECONDARY OUTCOMES:
Salivary Ductal Visibility | One year after completion of IMRT on last enrolled patient
  Correlation between mean dose to individual salivary gland ducts and post-treatment visibility scores
Salivary Gland Volume | One year after completion of IMRT on last enrolled patient
  Correlation between mean dose to individual salivary gland ducts and post-treatment salivary gland volume
Salivary Secretion Rate | One year after completion of IMRT on last enrolled patient
  Correlation between mean dose to individual salivary gland ducts and post-treatment saliva secretion rate
Salivary Secretion Recovery | One year after completion of IMRT on last enrolled patient
  Comparison of salivary secretion recovery rate after IMRT with salivary ductal sparing compared to current literature, particularly when irradiated glands exceed conventional dose constraints

CONTACTS AND LOCATIONS:
Overall Officials: David V. Fried, PhD, Principal Investigator — University of North Carolina at Chapel Hill, Department of Radiation Oncology
Locations (1):
- University of North Carolina at Chapel Hill, Department of Radiation Oncology, Chapel Hill, North Carolina, United States